CLINICAL TRIAL: NCT06256952
Title: SFB TRR 265: Losing and Regaining Control Over Drug Intake B03: Role of Pavlovian Mechanisms for Control Over Substance Use WP2: Effects of Social Isolation on PIT in AUD
Brief Title: Effect of Social Isolation on the Role of Pavlovian Mechanisms for Control Over Alcohol Use
Acronym: ReCoDe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Heidelberg University (Other); Zentralinstitut für Seelische Gesundheit Mannheim (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Andreas Heinz, Prof., MD, PhD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 40217046122
Record Dates: First submitted 2024-01-11; First posted 2024-02-13 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder; Alcoholism; Stress Reaction; Ostracism; Substance Use Disorders
Keywords: Substance use disorder (SUD); Alcohol use disorder (AUD); General and outcome-specific Pavlovian to instrumental transfer; Social exclusion; Humans; Surveys and Questionnaires; Reward; Cues
MeSH Terms: conditions — Alcoholism; Fractures, Stress; Ostracism; Substance-Related Disorders; Social Isolation

STUDY DESIGN:
Intervention Model Description: The study employs a within-group design. The participants of each group (AUD and HC) attend two consecutive sessions (one a day), and on each of these days, they engage in the Cyberball Experiment before undertaking the PIT Task. Within the Cyberball Experiment, participants are randomly assigned to either partial exclusion or inclusion on the first day. On the second consecutive day, they undergo the condition they did not experience previously.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (HC) - exclusion first (Experimental): Healthy participants without SUD Cyberball: Exclusion Day 1; Cyberball: Inclusion Day 2
  Interventions: Behavioral: PIT paradigm; Behavioral: social exclusion (Cyberball task); Diagnostic Test: Saliva samples; Diagnostic Test: basic psychological assessment; Diagnostic Test: pre and post cyberball task; Diagnostic Test: VAS; Diagnostic Test: after cyberball task; Behavioral: social inclusion (Cyberball task)
- Control (HC) - inclusion first (Experimental): Healthy participants without SUD Cyberball: Inclusion Day 1; Cyberball: Exclusion Day 2
  Interventions: Behavioral: PIT paradigm; Behavioral: social exclusion (Cyberball task); Diagnostic Test: Saliva samples; Diagnostic Test: basic psychological assessment; Diagnostic Test: pre and post cyberball task; Diagnostic Test: VAS; Diagnostic Test: after cyberball task; Behavioral: social inclusion (Cyberball task)
- Moderate to sever alcohol users (AUD) - exclusion first (Experimental): Participants with alcohol use disorder (moderate to severe if no withdrawal symptoms) and no other substance use disorder (SUD) Cyberball: Exclusion Day 1; Cyberball: Inclusion Day 2
  Interventions: Behavioral: PIT paradigm; Behavioral: social exclusion (Cyberball task); Diagnostic Test: Saliva samples; Diagnostic Test: basic psychological assessment; Diagnostic Test: pre and post cyberball task; Diagnostic Test: VAS; Diagnostic Test: after cyberball task; Behavioral: social inclusion (Cyberball task)
- Moderate to sever alcohol users (AUD) - inclusion first (Experimental): Participants with alcohol use disorder (moderate to severe if no withdrawal symptoms) and no other substance use disorder (SUD) Cyberball: Inclusion Day 1; Cyberball: Exclusion Day 2
  Interventions: Behavioral: PIT paradigm; Behavioral: social exclusion (Cyberball task); Diagnostic Test: Saliva samples; Diagnostic Test: basic psychological assessment; Diagnostic Test: pre and post cyberball task; Diagnostic Test: VAS; Diagnostic Test: after cyberball task; Behavioral: social inclusion (Cyberball task)

INTERVENTIONS:
Behavioral: PIT paradigm — The paradigm consists of four parts:
  In the first part, an instrumental learning task is completed in which subjects must learn which stimuli require a response and which do not. In the second part, a classical (Pavlovian) conditioning task is then completed in which subjects learn by passive viewing which stimuli are associated with certain amounts of money. The third part measures to which instrumental responses (learned in Part 1) are modulated by the presentation of the classically conditioned stimuli (learned in Part 2). At the same time drug-associated stimuli are presented in the background measuring to which extent they conflict with the learned instrumental behavior. In the last part, query trials are implemented in which the participants have to choose between two pictures to assess the relative cue value.
Behavioral: social exclusion (Cyberball task) — Social exclusion will be assessed using the cyberball paradigm: subjects will play an online game tossing a ball to each other with two more virtual co-players. Using a cover story, we make subjects believe that the co-players really exist and that they play a live online game. During social exclusion, subjects will be systematically excluded by one co-player, and during social inclusion, ball tosses will be balanced between all three players.
Diagnostic Test: Saliva samples — Assessing acute stress effects in AUD and HC subjects
Diagnostic Test: basic psychological assessment — * Sociodemographics
  * ASSIST
  * Quantity Frequency: Alcohol, tobacco/e-cigarette, Cannabis & other illegal drugs
  * SCID: AUD criteria and tabak use disorder life time and last year & acute depressive symptoms & symptoms for Mania and psychotic disorder
  * Edinburgh Handedness Inventory (EHI)
  * Fagerström Test for Nicotine depend (FTND)
  * Barratt Impulsiveness Scale - Kurzversion (BIS-15)
  * Allgemeine Depressionsskala (ADS)
  * State-Trait-Anxiety Inventory (STAI-T)
  * Alcohol Use Disorders Identification Test (AUDIT)
  * Cannabis Use Disorder Identification Test (CUDIT)
  * CAS -A (Alkohol)
  * Fragebogen zur Sozialen Unterstützung (F-SozU K-14)
  * Oslo-3-Items-Social-Support Scale
  * Social Skills Rating System (SSRS)
  * Trier Inventory for chronic stress (TICS)
  * Rejection Sensitivity Questionnaires (RSQ-9)
  * Need to belong scale (NTBS)
  * Fragebogen zu Gedanken und Gefühlen (FGG-14)
  * Internationale Trauma Questionnaire (ITQ)
  * Zahlen-Symbol-Test (DST)
  * Wortschatztest (verbal intelligence)
Diagnostic Test: pre and post cyberball task — Positive and Negative Affect Schedule(PANAS)
Diagnostic Test: VAS — subjective arousal, subjective stress, valence, perceived ostracisms/loneliness
Diagnostic Test: after cyberball task — * Need Threat Scale
  * Manipulation check (VAS scale)
Behavioral: social inclusion (Cyberball task) — Social inclusion will be assessed using the cyberball paradigm: subjects will play an online game tossing a ball to each other with two more virtual co-players. Using a cover story, we make subjects believe that the co-players really exist and that they play a live online game. During social inclusion, ball tosses will be balanced between all three players.

SUMMARY:
During the first funding period (1st FP) we investigated the impact of acute and chronic stress (Trier Social Stress Test, TSST) on Pavlovian-to-instrumental transfer (PIT). Moreover, we developed a novel full transfer task that allows assessing both general and specific PIT to investigate whether specific PIT differs between alcohol use disorder (AUD) and control subjects. We found that our online version of TSST induced stress and thereby amplified PIT effects in participants. Preliminary analyses of the full transfer task indicate that AUD participants exhibit a stronger specific PIT effect compared to controls. Based on these findings, we want to assess the following aim for this study:

Investigate the effect of experimentally induced social exclusion on alcohol-specific and general PIT effects in AUD and control participants.

DETAILED DESCRIPTION:
The projects research aim:

The investigators will examine how an experimentally induced social exclusion by the Cyberball task is associated with alcohol specific and general PIT effects by using the newly developed full transfer task from 1st funding period in AUD vs. HCs.

The investigators will use the newly developed full PIT paradigm to examine the modifying effect of experimentally induced social exclusion stress on alcohol-specific and general PIT effects. While using the Trier Social Stress Test in the 1st FP, the investigators now want to go one step further by including social exclusion/ostracism to the stress component, which has not been studied in association with PIT effects yet. The investigators here want to shed light on possible underlying mechanisms which can lead to a promotion of alcohol-seeking by alcohol-stimuli in situations of social exclusion.

Participants (50 AUD and 50 HC) will be assessed at two time points, once after experimentally induced social exclusion and once after social inclusion in a fully balanced, cross-over within-subject design. Subjects will play an online game tossing a ball to each other with two more virtual co-players (Cyberball). Using a cover story, we make subjects believe that the co-players really exist and that they play a live online game. During social exclusion, subjects will be systematically excluded by one co-player (partial exclusion), and during social inclusion, ball tosses will be balanced between all three players. Cyberball usually induces feelings of social isolation and altered behavioral reactions in the subject, which the investigators want to assess by analyzing ball tossing behavior over time, as well as physiological and subjective measures (concentration of cortisol in saliva, heart rate variability and emotions questionnaires, such as the Need to Belong Scale, Rejection Sensitivity Questionnaire, Need threat scale and Positive and Negative Affect Schedule pre and post Cyberball game and after PIT). After the Cyberball experiment, subjects will undergo the transfer part of the full PIT task (using a parallel version at one of the two days in a randomized order).

Hypothesis 1a:

Social exclusion will lead to a stronger stress hormone response (concentration of cortisol in saliva), lower heart rate variability and a stronger general PIT effect compared to social inclusion (main effect social exclusion intervention on PIT).

Hypothesis 1b:

Stronger social exclusion effects in AUD subjects compared to controls will lead to stronger PIT effects compared to social inclusion (interaction effect between group and stress intervention on PIT), especially for alcohol-specific PIT.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18-65 years of age,
* AUD subjects: meet 4 or more criteria for DSM-5 alcohol-use disorder (not requiring withdrawal as assessed by an independent psychiatrist),
* Currently using alcohol without a desire for abstinence,
* Ability to consent to the study and complete the questionnaires.
* Sufficient language skills: German
* Availability between 3pm-6pm on 2 consecutive days,
* existing health insurance

Exclusion Criteria:

* Lifetime diagnosis according to DMS-5 for a: Bipolar disorder, schizophrenia, schizophrenia spectrum disorder, substance dependence except for alcohol, nicotine, cannabis, and/or methamphetamine
* Currently meeting DSM-5 diagnostic criteria for depressive episode, suicidal ideation,
* History of traumatic brain injury or severe neurological disease (such as dementia, Parkinson's disease, multiple sclerosis)
* Pregnancy or breastfeeding,
* Ingestion of medications known to interact with the CNS in the 10-day period prior to study participation or less than 4 half-lives after last ingestion (rapid urine test),
* Color vision deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral full-lever specific and general PIT (parallel version) effect day one | Day 1
  Specific:
  Average percentage of alcohol choice difference during the presentation of alcohol or non-alcohol pavlovian background.
  General:
  Differences in number of button presses during the presentation of positive (+10 Euro) and negative (-10 Euro) pavlovian backgrounds.
Behavioral full-lever specific and general PIT (parallel version) effect day two | Day 2
  Specific:
  Average percentage of alcohol choice difference during the presentation of alcohol or non-alcohol pavlovian background.
  General:
  Differences in number of button presses during the presentation of positive (+10 Euro) and negative (-10 Euro) pavlovian backgrounds.
Social exclusion/inclusion induced using Cyberball Game | Day 1
  experimentally-induced social exclusion stress by using the cyberball paradigm: Subjects will play an online game tossing a ball to each other with two more virtual co-players. Using a cover story, we make subjects believe that the co-players really exist and that they play a live online game. During social exclusion, subjects will be systematically excluded by one co-player (partial exclusion), and during social inclusion, ball tosses will be balanced between all three players. Effects of the Cyberball manipulation (social exclusion/inclusion) will be assessed via ratings in Positive and Negative Affect Scale (PANAS) and Need-Threat-Scale (NTS).
Social exclusion/inclusion induced using Cyberball Game | Day 2
  experimentally-induced social exclusion stress by using the cyberball paradigm: Subjects will play an online game tossing a ball to each other with two more virtual co-players. Using a cover story, we make subjects believe that the co-players really exist and that they play a live online game. During social exclusion, subjects will be systematically excluded by one co-player (partial exclusion), and during social inclusion, ball tosses will be balanced between all three players. Effects of the Cyberball manipulation (social exclusion/inclusion) will be assessed via ratings in Positive and Negative Affect Scale (PANAS) and Need-Threat-Scale (NTS).

SECONDARY OUTCOMES:
Concentration of cortisol in saliva | Day 1 and Day 2
  [Time Frame: Assessment before, during and after Cyberball game (T1: arrival of subject), T2: right before Cyberball game, T3: right after Cyberball game, T4: after PIT part 3 and T5: at the end of testing day)]
Positive and Negative Affect Schedule (PANAS) | Baseline and after Cyberball Experiment on Day 1 and Day 2
  Scale 1-5, for PA (positive affect) and NA (negative affect) higher scores indicate higher positive and negative affect
Need Threat Scale (NTS) | After Cyberball Experiment on Day 1 and Day 2
  Scale from 1 to 5, high scores indicate high needs in Belonging, Control, Meaningful existence and self-esteem
Heart rate variability | At baseline 5 min AND During experimental part (social inclusion or exclusion) 5 min Day 1 and Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- Charite - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Roayaee M, Rahman RA, Danziger M, Tudge L, Daedelow LS, Heinz A, Wustenberg T. [The others and I: How social interactions change the perception of other persons. The Cyberball paradigm and its indications in the migration context]. Fortschr Neurol Psychiatr. 2020 Feb;88(2):109-117. doi: 10.1055/a-1033-7304. Epub 2020 Feb 26. German. PMID 32102102
- [Background] Staebler K, Helbing E, Rosenbach C, Renneberg B. Rejection sensitivity and borderline personality disorder. Clin Psychol Psychother. 2011 Jul-Aug;18(4):275-83. doi: 10.1002/cpp.705. Epub 2010 May 25. PMID 21110407